CLINICAL TRIAL: NCT04918810
Title: A Phase II Trial of Biomarker-driven Intermittent Docetaxel in Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Biomarker-driven Intermittent Docetaxel in Metastatic Castration-resistant Prostate Cancer
Acronym: GUIDE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment lower than expected. The proportion of patients with mGSTPi undetectable prior to chemo. was significantly higher than anticipated. Decision made to close due to insufficient patient numbers to able to obtain meaningful data collection.
Sponsor: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP 1903
Record Dates: First submitted 2021-05-26; First posted 2021-06-09 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Castration Resistant Prostatic Cancer
Keywords: mGSTPi
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1: Intermittent docetaxel treatment (Experimental): suspend docetaxel prior to cycle 4, recommencement based on mGSTP1 monitoring
  Interventions: Drug: Docetaxel intermittent

INTERVENTIONS:
Drug: Docetaxel intermittent — After 3 or 4 cycles of docetaxel chemotherapy (75mg/m^2 every 21 days or 50mg/m^2 every 14 days) in combination with an undetectable mGSTP1 level, patients will stop docetaxel treatment. Plasma mGSTP1 is measured every 21 days or 28 days (depending on Docetaxel regimen) and docetaxel treatment will be recommenced if it mGSTP1 becomes detectable again.

SUMMARY:
The purpose of this study is to see if a prostate cancer marker in the blood (mGSTP1) can be used to guide chemotherapy treatment. Based on the level of this blood marker, some people may be able to have breaks in treatment rather than having chemotherapy continuously which is the current standard of care. This study will tell us if having these treatment breaks guided by mGSTP1 can improve how people feel during treatment while still treating the prostate cancer effectively.

Docetaxel is a chemotherapy drug that is approved to treat prostate cancer and has been used for many years to treat prostate cancer like yours. Your doctor has already discussed this with you and you have both agreed that docetaxel is the best treatment for you to have at this time. You will have already started this chemotherapeutic treatment with docetaxel.

ELIGIBILITY:
PRESCREENING INCLUSION CRITERIA

1. Patient has provided written informed consent using the GUIDE pre-screening PICF
2. Age ≥ 18 years at the time of pre-screening consent
3. Males with metastatic castration-resistant prostate cancer (as per PCWG3) AND are planned to commence docetaxel chemotherapy
4. WHO Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Appendix 1)
5. Histological confirmation of prostate cancer
6. Patients must have adequate bone marrow and hepatic function within 14 days prior Cycle 1 day 1:

   * Haemoglobin ≥ 90 g/L independent of transfusions (no red blood cell transfusion in last 4 weeks)
   * Platelets ≥ 100 x 109/L
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * Alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) ≤ 2.5 x ULN
7. Willing and able to comply with all pre-screening study requirements, including blood tests for mGSTP1 analysis before and during docetaxel treatment

PRESCREENING EXCLUSION CRITERIA

1. Prior docetaxel or cabazitaxel chemotherapy for castration-resistant prostate cancer
2. Prior docetaxel in the castration sensitive prostate cancer setting within the previous 2 years
3. Known hypersensitivity to docetaxel or its excipients
4. Concurrent illness, including severe infection that may jeopardise the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety
5. Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol

MAIN SCREENING INCLUSION CRITERIA

1. Patient has provided written informed consent for the main GUIDE study PICF
2. Patient has a detectable plasma mGSTP1 deoxyribonucleic acid (DNA) as measured by central laboratory at prescreening prior to commencing first cycle of docetaxel chemotherapy
3. Patient has commenced 3 cycles of docetaxel
4. Patient has undetectable plasma mGSTP1 DNA as measured by central laboratory from blood taken prior to the third cycle of docetaxel
5. Patient is willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments.

MAIN SCREENING EXCCLUSION CRITERIA

1. Known hypersensitivity to docetaxel or its excipients
2. Concurrent illness, including severe infection that may jeopardise the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety
3. Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol
4. Progressive disease by RECIST 1.1 within the first 3 cycles of docetaxel

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Radiographic progression free survival (rPFS) | From enrollment until last patient has completed 2 years in follow up, on average 3.5 years
  Radiographic progression free survival (rPFS) is defined as the time from enrollment (i.e. prior to cycle 4), the date of first documented progression on imaging by site investigator (PCWG3 criteria for bone lesions and RECIST 1.1 for soft tissue lesions) or death due to any cause.

SECONDARY OUTCOMES:
Time on treatment holidays | From enrollment until last patient has completed 2 years in follow up, on average 3.5 years
  Time on treatment holidays is defined as the total length of time patients on the intermittent docetaxel spend off docetaxel within the treatment period i.e. prior to permanent treatment discontinuation
Overall treatment safety | From the date of signing consent on the Main study until 90 days after the last day of protocol treatment, on average 3.5 years
  Incidence and severity of adverse events (AEs) using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.
Overall survival | From enrollment until last patient has completed 2 years in follow up, on average 3.5 years
  Overall survival is defined as the time from enrollment to the date of death due to any cause
Overall quality of life | From enrollment until last patient has completed 2 years in follow up, on average 3.5 years
  Quality of Life using the EORTC QLQ-C30 (European Organisation for Research on Treatment of Cancer - Quality of Life Questionnaire for cancer patients) instrument.
  The instrument uses 28 questions about overall quality of life with each question answerable using a scale from 1 (not at all) to 4 (very much). Overall scores can be from a minimum of 28 indicating a better quality of life and higher scores with a maximum of 112 indicating lower overall quality of life.
  The questionnaire also has two summary questions which asks participants to rank 1) overall health and 2) overall quality of life on scale of from 1, very poor, to 7, excellent.
Fatigue | From enrollment until last patient has completed 2 years in follow up, on average 3.5 years
  Fatigue, using the EORTC FA-12 (European Organisation for Research on Treatment of Cancer - Fatigue) instrument.
  This instrument uses 12 questions for participants about fatigue with each question answerable on a scale of 1 (not at all) to 4 (Very Much) to a maximum score of 48 indicating worse overall self-rated fatigue.
Fear of progression | From enrollment until last patient has completed 2 years in follow up, on average 3.5 years
  Fear of progression using the short FOP12 (Fear of Progression) instrument.
  This instrument uses 12 questions about participant's own Fear of Progression with each question answerable using a scale from "Never" to "very often" with lower scores indicating a better outcome.
Patient reported adverse events | From enrollment until last patient has completed 2 years in follow up, on average 3.5 years
  Patient reported adverse events using the patient reported modified PRO-CTCAE instrument
Frequency of health resource utilisation | From time of consent until End of Study, on average 3.5 years
  To compare resource use associated with mGSTP1 directed therapy. Will be measured from trial based eCRFs and will include frequency of mGSTP1 testing, use of docetaxel and corticosteroids, pathology tests and imaging.
  People participating in the GUIDE study will be consented for access to their Medicare claims data providing information on outpatient use of PBS listed therapies (such as those for metastatic bone disease) and Medicare services (such as outpatient clinician services)
Overall cost associated with treatment | From time of consent until End of Study, on average 3.5 years
  To compare costs associated with treatment. Will be reported by type of health care used and the total cost of health care used over the period of the trial and follow-up.
  Market prices will be applied to items of resource use to estimate costs.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Mahon, Principal Investigator — Chris Obrien Lifehouse
Locations (8):
- Australia (8):
  - Border Medical Oncology Research Unit / The Border Cancer Hospital, Albury, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Dubbo Base Hospital, Dubbo, New South Wales
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Frankston Hospital-Peninsula Health, Frankston, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - LaTrobe Regional Hospital, Traralgon, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ANZUP website — https://www.anzup.org.au/